CLINICAL TRIAL: NCT06513377
Title: Evaluating and Monitoring Physical Fatigue While Performing Functional Activities
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vrije Universiteit Brussel (Other)
Responsible Party: Principal Investigator, David Beckwee, Principal Investigator, Vrije Universiteit Brussel
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: RevalExo2
Record Dates: First submitted 2024-06-25; First posted 2024-07-22 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2025-09

CONDITIONS: Stroke; Sarcopenia; Fatigue
MeSH Terms: conditions — Stroke; Sarcopenia; Fatigue

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- People post-stroke (Experimental): The intervention includes a stress test that induces progressive feelings of fatigue.
  Interventions: Other: Performance test
- Older adults with sarcopenia (Experimental): The intervention includes a stress test that induces progressive feelings of fatigue.
  Interventions: Other: Performance test
- Healthy individuals (Experimental): The intervention includes a stress test that induces progressive feelings of fatigue.
  Interventions: Other: Performance test

INTERVENTIONS:
Other: Performance test — The participant will be asked to execute a protocol in the movement lab that induces progressive feelings of fatigue. This protocol includes a sequence of relevant functional activities, such as stair walking, slope walking, crouching, walking different path shapes. During this execution the Ratings of Perceived Exertion will be questioned, and simultaneously physiological and movement data will be collected.

SUMMARY:
Fatigue is a critical health parameter in older adults and stroke patients and is associated with negative health outcomes. Current assessment tools predominantly focus on walking related fatigue, neglecting other activities of daily living (ADLs). This study aims to fill this gap by developing a standardized, laboratory-based fatigue protocol that includes a broader range of ADLs, providing a more comprehensive fatigue assessment that's in line with the WHO vision of healthy ageing.

The aim of this study is to evaluate a lab-based fatigue protocol and to unravel the relationship between physiological or movement data and perceived fatigue.

Participants will take part in three separate measurement moments, during which they will execute a performance task that induces fatigue. In addition, relevant sensors will be used to collect meaningful data.

ELIGIBILITY:
Stroke survivors:

Inclusion Criteria:

* > 18 years old
* ≥ 3 months ago stroke diagnosis
* FAC levels 3-5

Exclusion Criteria:

* Severe problems with speech or memory which prevents the participant to understand or follow instruction
* Co-morbidities that could influence the task execution and collected data

Older adults with sarcopenia:

Inclusion:

* > 65 years old
* Grip strength: < 27 kg (man) or < 16 kg (woman)
* Be mobile independently

Exclusion:

* Severe problems with speech or memory which prevents the participant to understand or follow instruction
* Co-morbidities that could influence the task execution and collected data

Healthy individuals:

Inclusion:

* > 18 years old
* Healthy physical and medical condition

Exclusion:

* Physical injury or disorder that doesn't allow good physical performance

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2025-03-20 (Actual); Primary Completion 2025-10-15 (Actual); Study Completion 2025-10-15 (Actual)

PRIMARY OUTCOMES:
Changes in the Ratings of Perceived Exertion throughout the protocol execution | Collected during all measurement moments (2-12 weeks).
  The subjective feelings of fatigue will be evaluated through the Ratings of Perceived Exertion. This will be expressed verbally by the participant throughout the execution of the protocol.

SECONDARY OUTCOMES:
Changes in muscle activity throughout the protocol execution | Collected during all measurement moments (2-12 weeks).
  Muscle activity data (EMG) will be collected continuously throughout the protocol execution. Data acquisition will occur in a synchronized manner.
Changes in heart rate (variability) throughout the protocol execution | Collected during all measurement moments (2-12 weeks).
  Cardiorespiratory data (Heart rate) will be collected continuously throughout the protocol execution. Data acquisition will occur in a synchronized manner.
Changes in oxygen saturation throughout the protocol execution | Collected during all measurement moments (2-12 weeks).
  Oxygen saturation data will be collected continuously throughout the protocol execution. Data acquisition will occur in a synchronized manner.
Changes in electrodermal activity throughout the protocol execution | Collected during all measurement moments (2-12 weeks).
  Electrodermal activity data will be collected continuously throughout the protocol execution. Data acquisition will occur in a synchronized manner.
Changes in muscle force myography throughout the protocol execution | Collected during all measurement moments (2-12 weeks).
  Muscle force myography data will be collected continuously throughout the protocol execution. Data acquisition will occur in a synchronized manner.
Changes in skin temperature throughout the protocol execution | Collected during all measurement moments (2-12 weeks).
  Skin temperature data (degrees Celsius) will be collected continuously throughout the protocol execution. Data acquisition will occur in a synchronized manner.
Changes in motion data throughout the protocol execution | Collected during all measurement moments (2-12 weeks).
  IMU data will be collected continuously throughout the protocol execution. Data acquisition will occur in a synchronized manner.
Changes in plantar pressure throughout the protocol execution | Collected during all measurement moments (2-12 weeks).
  Plantar pressure distribution data will be collected continuously throughout the protocol execution. Data acquisition will occur in a synchronized manner.
Changes in gaze patter throughout the protocol execution | Collected during all measurement moments (2-12 weeks).
  Eye tracking data will be collected continuously throughout the protocol execution. Data acquisition will occur in a synchronized manner.
Changes in joint angles throughout the protocol execution | Collected during all measurement moments (2-12 weeks).
  Kinematic data (degrees) will be collected continuously throughout the protocol execution. Data acquisition will occur in a synchronized manner.

CONTACTS AND LOCATIONS:
Locations (1):
- Brubotics Rehabilitation Research Center, Jette, Brussels Capital, Belgium